CLINICAL TRIAL: NCT02497846
Title: Feasibility and Acceptability of a TEOSYAL® PureSense Redensity [I] Injection Using MicronJet® Needle in the Treatment of Crow's Feet Wrinkles
Brief Title: TEOSYAL® PureSense Redensity [I] Injection Using MicronJet® Needle in the Treatment of Crow's Feet Wrinkles
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Teoxane SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TEO-R1-1404
Record Dates: First submitted 2015-05-18; First posted 2015-07-15 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2015-05

CONDITIONS: Crow's Feet Wrinkles
Keywords: Hyaluronic acid; MiconJet needle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TEOSYAL® PureSense Redensity [I]/MicronJet® (Experimental): injection of the acid hyaluronic gel with lidocaine as an anesthetic and a "dermo-restructuring complex (including 8 amino acids , 3 antioxidants Acid, vitamin B6 and 2 minerals).
  Product will be injected in a unique device group:
  * in crow's feet in order to cover the zone to be treated. Quantity of product injected will be determined by the injector and noted (up to 1 ml by side). A subject can be injected in the left or/and right side.
  * using a MicronJet microneedle for the superficial wrinkles.
  Interventions: Device: TEOSYAL® PureSense Redensity [I]/MicronJet®

INTERVENTIONS:
Device: TEOSYAL® PureSense Redensity [I]/MicronJet® — According the instruction of use, 3 injections of TEOSYAL® PureSense Redensity [I]will be performed all the 3 weeks. The used needle will be the MicronJet® microneedles for product injection. And the last visit (of control) will be performed 3 weeks after the last injection.

SUMMARY:
The purpose of this study is to evaluate the feasibility and acceptability of a TEOSYAL® PureSense Redensity [I] injection using MicronJet® needle in the treatment of crow's feet wrinkles.

It is a monocentric, open-blind, prospective, pilot study. 3 injections sessions spaced with an interval of 3 weeks. The last visit will be performed 3 weeks after the last injection.

Only, one group of 15 healthy volunteers will be included.

DETAILED DESCRIPTION:
TEOSYAL® PureSense Redensity [I] is a viscoelastic gel of non-cross-linked hyaluronic acid that is sterile, non pyrogenic, colourless and of non-animal origin and contains 0.3% by mass of lidocaine hydrochloride, for its anaesthetic properties. Each box contains two syringes pre-filled with Teosyal® PureSense Redensity I. The volume of each syringe is shown on the cardboard box as well as on each syringe. Teosyal® PureSense Redensity I is indicated for the prevention of wrinkles and rehydration of the neck, neckline, face and in particular the crow's feet wrinkles.

The MicronJet® needle is a 3 micro-needle (0.6 mm of length) device that is mounted on a standard syringe in the same manner as a conventional needle. The MicronJet® needle is used to inject liquid substances, allowing for controlled intradermal delivery in any procedure which requires administration of substances to the dermal compartment.

For the first time, the TEOSYAL® PureSense Redensity [I] will be injected using the medical device MicronJet® in the superficial wrinkles.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer (desiring an aesthetic improvement of crow's feet area).
* Crow's feet score between 3 to 5 on both sides.
* Psychologically able to understand the study related information (For example, it will be difficult to include a foreigner who does not speak French, unaccompanied by a translator or subject who can't read the information note and the volunteer diary).
* Having given his informed consent.
* Female subjects of childbearing potential should use a medically accepted contraceptive regimen (for example, hormonal contraception, intrauterine contraceptive device or surgical sterilization…), during all the study and at least 1 month after the study end.

Exclusion Criteria:

* Pregnant or nursing woman or planning a pregnancy during the study (according to the product IFU).
* Volunteer having a previous history of cutaneous cancer or all others type of cancer. (to verify that the volunteer is healthy)
* Suffering from a serious or progressive diseases, which, put the subject at undue risk (as for example diabetes, auto-immune pathology, cardiac pathologies, hepatic deficiency, epilepsy )(to verify that the volunteer is healthy)
* With scars, infection, or other pathology on the injection sites. (as rosacea, herpes, acne, blotches on the injection sites. (the product injection can't be performed on a damaged skin and the wrinkles can be seen by the investigator - according to the product IFU)
* With active skin disease within 6 months prior to study entry. (according to the product IFU)
* With severe rheumatism fever.
* Predisposed to keloidosis (itchy skin or skin rash and hives) or hypertrophic scarring. (
* With a known allergy to one of the ingredients of the tested products (as hyaluronic acid hypersensitivity or lidocaine or local anesthetic: 70° Alcohol or Chlorhexidine allergy). (according to the product IFU)
* With multiple allergies or anaphylactic shock history. (according to the product IFU)
* With coagulation troubles, abnormal bleeding as hemophiliac or von Willebrand disease.
* Under an anti-coagulant treatment in the 2 weeks preceding the study.
* Under >30,000 IU/day oral vitamin E in the 1 week preceding the study.
* Under corticosteroids in the 2 weeks preceding the study and used in the severe allergy treatment.
* Under interferon in the 1 month preceding the study and used for antiinfectious or antioncogene proprieties.
* Having an aspirin (ASA - Acetyl Salicylic Acid) or a non-steroidal anti-inflammatory treatment in the last 15 days (the subject can still be bled easily).
* Having a peeling, laser or ultrasound-based treatment. (according to the product IFU)
* Having any medication which may interfere, at the interpretation of the investigator, with the study objectives in term of efficacy and safety tolerance (currently, the interactions with an other HA product are not tested, it is not possible to inject Teosyal® PureSense Redensity I into sites where other filling implants are present - according to the product IFU).
* Suspected to be non-compliant according to the investigator's judgment (for example, a subject for which the investigator knows that he cannot come to all the visits in reason of holidays or moving, can be not include in this study)
* Enrolled in another clinical trial or being in an exclusion period for a previous study.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-05; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Crow's feet responder for the feasibility outcome | Day 63 (end of study)
  The crow's feet responder is defined as a crow's feet score with at least one grade of improvement between D0 and D63. As the subject can be treated on each side, each subject can give two answers.

SECONDARY OUTCOMES:
Subject satisfaction for acceptability outcome | at Day 0, Day 21, D42 and D63 (end of study visit)
  5-grade Likert scale
Pain evaluated by the subject | at Day 0, Day 21 and D42
  Subjective visual analogue scale (0 to 10 cm)

OTHER OUTCOMES:
Adverse event | From Day 0 to Day 63 (end of study)
Local reactions collected by the subject | at Day 0, Day 21 and D42
  Local reactions collected by the subject on a 14-day subject diary
Change from Baseline of crow's feet scale (Aesthetic Improvement) for efficacy Measurement | at Day 21, Day 42 and Day 63 (end of study visit)
  7-grade scale
Global Aesthetic Improvement scale for efficacy measurement | at Day 21, Day 42 and Day 63 (end of study visit)
  5 grade likert scale
Product leakage at the skin area, in comparison with a classic needle | at Day 63 (end of study visit)
  4-grade scale
Pain sensation at the insertion, in comparison with a classic needle | at Day 63 (end of study visit)
  4-grade scale

CONTACTS AND LOCATIONS:
Locations (1):
- Docteur MICHEELS, Geneva, Switzerland